CLINICAL TRIAL: NCT04498091
Title: EPIdemiological Approaches to the Cardiovascular Consequences of COVID-19
Acronym: EPI CV COVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Zeller AOIc 2020
Record Dates: First submitted 2020-08-03; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A: Type 2 MI with COVID-19
  Interventions: Biological: Biological data; Other: Clinical data
- B: Type 2 without COVID-19
  Interventions: Biological: Biological data; Other: Clinical data
- C: Type 2 MI with pneumonia without COVID-19
  Interventions: Biological: Biological data; Other: Clinical data
- D: Type 2 MI without pneumonia and without COVID-19
  Interventions: Biological: Biological data; Other: Clinical data

INTERVENTIONS:
Biological: Biological data — Biological data
Other: Clinical data — Clinical data

SUMMARY:
The COVID-19 pandemic highlights the importance of the prognosis of co-morbidities, such as coronary artery disease, which significantly increase the risk of mortality in patients infected with SARS-CoV2. Investigators have recently studied the complex links between respiratory infections, particularly pneumonia, and type 2 myocardial infarction (MI) in many respects. The etiology of type 2 MI is based on an imbalance of myocardial oxygen supply/need in the absence of rupture/erosion of atheromatous plaques. Based on the RICO survey data, the investigators investigated whether COVID-19-related sepsis and/or respiratory failure could be an underlying mechanism of MI2.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized for a type 2 MI in CCU from CHU Dijon Bourgogne With or without pneumonia
* patients hospitalized for a type 2 MI in CCU from CHU Dijon Bourgogne With or without COVID 19

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute type 2 MI
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Characterizing type 2 myocardial infarction associated with CoV-2 SARS infection | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France